CLINICAL TRIAL: NCT07205055
Title: Effect of Video-Based Diaper Dermatitis Care Education on Mothers' Knowledge Level and Dermatitis Severity: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Gunay Arslan, assistant professor, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: UU-SBF-GA-01
Record Dates: First submitted 2025-09-24; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Diaper Dermatitis; Diaper Rash; Diaper Dermatitis Healing
Keywords: mother; education; video; diaper dermatitis; napkin dermatitis; diaper rash
MeSH Terms: conditions — Diaper Rash

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study (Active Comparator): The severity of diaper dermatitis will be monitored by having the mothers in the study group watch a video training session. This will allow for the healing effect to be observed.
  Interventions: Other: video training
- CONTROL (No Intervention): NO APPLICATION WILL BE MADE

INTERVENTIONS:
Other: video training — No study in the literature has examined the effectiveness of video-based diaper dermatitis education.
  Arms: study

SUMMARY:
This study was conducted using a randomized controlled, pretest-posttest comparative experimental design to examine the effects of diaper dermatitis care training provided to primiparous mothers on mothers' knowledge and the severity of diaper dermatitis in infants aged 0-6 months. The study was conducted with a total of 74 primiparous mothers from June to September 2025. Participants were divided into intervention (n=37) and control (n=37) groups. The intervention group received video training on diaper dermatitis care.

DETAILED DESCRIPTION:
Purpose of Study This study aims to investigate the effects of video diaper dermatitis care training provided to primiparous mothers on diaper dermatitis severity scores and mothers' knowledge levels in 0-6 month-old infants.

Research Type This study is a randomized controlled, pretest-posttest comparative, experimental design to determine the effects of video diaper dermatitis care training provided to primiparous mothers on diaper dermatitis severity scores and mothers' knowledge levels in 0-6 month-old infants.

Place and Time of Study The study was conducted at a city hospital on the Anatolian side of Istanbul. The third floor of this hospital houses seven general pediatrics outpatient clinics, two pediatrics and infection clinics, and two pediatric hematology and oncology outpatient clinics. Services on the outpatient clinic floor include laboratory tests, imaging, health reports, patient admission procedures, well-child follow-up and examination, sick-child follow-up and examination, vaccination follow-up and referral, and lactation and relactation training. This hospital was selected because it is the researcher's affiliated institution and because of its diverse patient population.

The research was conducted between June and September 2025.Research Hypotheses H1: There is no significant difference between the pretest and posttest scores of the Mothers' Child Care Knowledge and Practice Level Assessment Form for the mothers in the control group.

H2: The posttest score of the Mothers' Child Care Knowledge and Practice Level Assessment Form for the mothers in the study group is higher than the pretest score.

H3: The posttest score of the Mothers' Child Care Knowledge and Practice Level Assessment Form for the mothers in the study group is higher than the control group.

H4: The final score of the Infant Uncomplicated Diaper Dermatitis Severity Rating Scale for the infants in the study group is lower than the control group.

H5: The final score of the Infant Uncomplicated Diaper Dermatitis Severity Rating Scale for the infants in the study group is lower than the pretest score.

Research Population and Sample A power analysis was conducted to determine the number of participants to be included in the study. The power of the test was calculated using the G*Power 3.1.9.2 program. In a similar study in the relevant literature, Nur Çelik (2023) calculated the effect size for dermatitis as 0.847. To exceed 95% power, a 5% significance level and an effect size of 0.847 required reaching 62 participants (df=60; t=1.671). Considering the high power of the test and the 20% loss, it was determined that a total of 74 participants (37 in each group) were needed. In the study, 74 mothers were divided into two groups. The first group (n=37 mothers) was the intervention group, which watched an educational video, and the second group (n=37 mothers) was the control group.

Randomized Study Seventy-four primiparous mothers and their infants, aged newborn-six months, who presented to the pediatric outpatient clinic, were registered on the CalculatorSoup website and divided into two groups. The numbers presented in Table 1 were obtained accordingly. Using random numbers generated based on the order of application, mothers and their babies were assigned to groups using a simple random sampling method. The sealed envelope method was used to determine which group the first case would be included in; envelopes were labeled "Intervention" and "Control" and sealed, and group assignment was made based on the contents of the envelope opened for the first case. Participants who declined to participate in the study were included in the first mother in the order. Verbal and written consent was obtained from the randomly assigned participants, and this process continued until the sample size was reached.

Inclusion Criteria for the Study

Infants aged 0-6 months and their mothers who applied to the child health clinic of the city hospital where the study would be conducted, Parents over 19 years of age, Volunteering for the study, Mothers having an only child, Having at least a primary school degree,

Exclusion Criteria for the Study

Infants with chronic diseases, Infants with dermatological or other allergic skin conditions, Having started complementary feeding, Being a healthcare professional, Mothers having a condition (physical, neurological, or mental) that prevents them from providing care, Those using diapers other than disposable diapers (free of perfume, phthalates, chlorine, dioxin, latex, or parabens).

Research Implementation Steps

Step 1: Research data were collected through face-to-face interviews. The study population consisted of mothers who applied to the pediatric outpatient clinic of the hospital where the study was conducted, met the research criteria, and volunteered to participate. Verbal and written consent was obtained from the mothers who agreed to participate in the study, and two separate groups were formed using a randomization method. Because participants who received the training might realize they were in the intervention group, the study will be conducted in an open-label, randomized manner. The randomization calculation, calculated via Calculatur.com, was provided to Keskin, the department secretary, and the researcher will not be aware of the intervention and control groups.

Step 2: Mothers in the experimental and control groups completed the "Mother and Baby Identification Form" and the "Mothers' Child Care Knowledge and Practice Level Assessment Form." The baby's diaper dermatitis was assessed at the bedside, and the "Uncomplicated Diaper Dermatitis Severity Assessment Scale (preliminary score)" was completed, and the pre-training severity score was recorded.

Step 3: Mothers in the experimental group watched a diaper dermatitis prevention and care video prepared by the researchers on the first day they arrived at the outpatient clinic and were enrolled in the study. The control group received no treatment. They were only instructed to follow their routine treatments as directed by their physician.

Step 4: In a survey conducted by Yıldız et al. (2023) with 217 pediatricians in 32 different provinces of Türkiye, 39.2% (n=85) of participants responded "7 days later" to the question, "After the initial evaluation, when would you recommend checking a patient with diaper dermatitis?" and 32.3% (n=70) recommended checking "3 days later" (Yıldız et al., 2023).

The mothers and their babies in the experimental and control groups were called to the hospital 7 days after their visit to the outpatient clinic. The "Mothers' Child Care Knowledge and Practice Level Assessment Form" was completed. The infant's diaper dermatitis was assessed at the bedside, and the "Uncomplicated Infant Diaper Dermatitis Severity Assessment Scale (final score)" was completed, and the severity score was recorded after the training.

Step 5: The study was concluded when the sample size was reached. Step 6: After the study was concluded, the mothers in the control group also watched the video training in accordance with ethical principles.

Limitations of the Study

The study was conducted only on mothers and their babies admitted to a single city hospital. The participants reflected specific socioeconomic and sociocultural characteristics, making it difficult to generalize nationwide.

Dependent and Independent Variables of the Study Independent Variables Sociodemographic Characteristics: Mother's age, education level, economic status, baby's gender, age, weight, height, baby's feeding habits, etc.

Video-based educational intervention Dependent Variables BSOBSS score AABBUDF score

Data Analysis of the Study Statistical Package for Social Sciences (SPSS) v27 was used for statistical analysis. Participant characteristics are presented using the number (n) and percentage (%), mean, standard deviation, minimum, and maximum values. Whether the control and intervention groups exhibited a conjugate structure in terms of descriptive characteristics was checked with chi-square analysis for categorical variables and independent groups t-test for numerical variables.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 0-6 months and their mothers who applied to the child health clinic of the city hospital where the study will be conducted,
* Parents over the age of 19,
* Volunteering for the study,
* The mother is an only child,
* Having at least a primary school degree,

Exclusion Criteria:

* Babies with chronic illnesses
* Babies with dermatological or other allergic skin conditions
* Being a healthcare professional
* Mothers with a medical condition (physical, neurological, or mental) that prevents them from providing care
* Those using diapers other than disposable diapers (free of perfume, phthalates, chlorine, dioxin, latex, or parabens)

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Primiparous mothers with babies aged 0-6 months
Enrollment: 74 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-18 (Actual)

PRIMARY OUTCOMES:
Mothers' Child Care Knowledge and Practice Level Form | 7 days
  The Mothers' Child Care Knowledge and Practice Level Assessment Form, prepared for use in the research process, was sent to 15 experts via e-mail to measure its content validity. Opinions were received from 10 experts, and these opinions were analyzed using appropriate methods. A three-item structure was used in the evaluation of the Mothers' Child Care Knowledge and Practice Level Assessment Form, which consists of 25 items: "item appropriate," "minor modifications needed," and "item not appropriate." Therefore, the Lawshe (1975) technique was utilized in the expert opinion analysis of the Mothers' Child Care Knowledge and Practice Level Assessment Form. The CVR and CGI values obtained as a result of the analysis are expected to be higher than the criterion value for the 10 experts, CGI=0.62 (Veneziano & Hooper, 1997). As a result of the analyses, it was determined that the CVR values for the items on the Mothers' Child Care Knowledge and Practice Level Assessment Form were in th

SECONDARY OUTCOMES:
Uncomplicated Diaper Dermatitis Severity Rating Scale in Infants | 7 DAYS
  The Uncomplicated Diaper Dermatitis Severity Assessment Scale (UCDDS) is a four-item scale developed by Buckley and colleagues in 2016. In the study in which the scale was developed, the Cronbach's alpha value was found to be 0.702 (Buckley et al., 2016). The Turkish adaptation of the scale was conducted by Keskin in 2019, and validity and reliability studies were also conducted. The Cronbach's alpha value was found to be 0.81 in the Turkish adaptation. The reliability coefficients of the items were reported as 0.73, 0.80, 0.78, and 0.79, respectively.
  Possible scores on the UCDDS range from 0 to 6. A higher total score indicates an increased severity of diaper dermatitis.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Lütfi Kırdar City Hospital, Istanbul, kartal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
If anyone wants to do any meta-analysis after the study is published, they can contact me via email.